CLINICAL TRIAL: NCT02556593
Title: IMRT Combined With Erlotinib Compared With Whole-brain Radiotherapy for EGFR Wild Type Non-small Cell Lung Cancer With 4-10 Brain Metastases
Brief Title: IMRT Combined With Erlotinib for EGFR Wild Type Non-small Cell Lung Cancer With 4-10 Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1009
Record Dates: First submitted 2015-09-19; First posted 2015-09-22 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Non-Small Cell Lung Carcinoma
Keywords: Non-Small Cell Lung Cancer; IMRT; erlotinib; whole-brain radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMRT & erlotinib (Experimental): Patients in experimental group receive IMRT and erlotinib: Daily IMRT(45Gy in 15 fractions) to the brain metastases with daily erlotinib(150mg.po) for three weeks
  Interventions: Radiation: IMRT; Drug: erlotinib
- whole-brain radiotherapy (Active Comparator): Patients in this group receive WBRT at 30Gy in 10 fractions
  Interventions: Radiation: WBRT

INTERVENTIONS:
Radiation: IMRT — Daily IMRT at 45 Gy in 15 fractions to brain metastases
  Arms: IMRT & erlotinib
Radiation: WBRT — 3DCRT at 30 Gy in 10 fractions to whole brain
  Arms: whole-brain radiotherapy
Drug: erlotinib — erlotinib 150mg daily
  Arms: IMRT & erlotinib

SUMMARY:
This study is to assess the efficacy of IMRT combined with erlotinib compared with whole-brain radiotherapy for EGFR wild type non-small cell lung cancer with 4-10 brain metastases.

DETAILED DESCRIPTION:
This study is to assess the efficacy of IMRT combined with erlotinib compared with whole-brain radiotherapy for EGFR wild type non-small cell lung cancer with 4-10 brain metastases.

All patients recruited will be randomly assigned into two groups. Patients in experimental group will receive daily IMRT at 45 Gy in 15 fractions to brain metastases, combined with daily erlotinib of 150mg for three weeks. Patients in control group will receive daily whole-brain radiotherapy at 30 Gy in 10 fractions.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed NSCLC and wild type EGFR
* 4-10 brain metastases on high quality CT scanning or MRI.
* No previous EGFR-TKI treatment.
* No previous brain radiotherapy.
* More than 4 weeks from last chemotherapy.
* Expected Survival of at least 2 months.
* KPS≥ 70
* RTOG RPA performance status 0-1
* Lab tests should meet these criteria: White blood cell count ≥3×10^9 /L;Platelet count≥100×10^9 /L;Total bilirubin 1.5 times or less the upper limits of normal (ULN); AST and ALT 1.5 times or less the ULN; Serum creatinine 1.5 times or less the ULN or creatinine clearance rate(CCR) greater than or equal to 60 ml/min.
* Pregnancy test (-)
* Be able to sign informed consent form.

Exclusion Criteria:

* With unstable systematical diseases (concluding acute infection, grade 4 hypertension, unstable angina pectoris, congestive heart failure, hepatopathy, nephropathy, metabolic diseases)
* With metastases on meninges.
* Taking antiepileptics (phenytoin sodium etc.) at the same time
* Unable to oral medication.
* Previous or recent another malignancy, except for nonmelanoma skin cancer or cervical cancer in situ

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
CNS progression free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Hui Liu, Guangdong, China

REFERENCES:
- [Background] Tsao MN, Lloyd N, Wong RK, Chow E, Rakovitch E, Laperriere N, Xu W, Sahgal A. Whole brain radiotherapy for the treatment of newly diagnosed multiple brain metastases. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD003869. doi: 10.1002/14651858.CD003869.pub3. PMID 22513917
- [Background] Pesce GA, Klingbiel D, Ribi K, Zouhair A, von Moos R, Schlaeppi M, Caspar CB, Fischer N, Anchisi S, Peters S, Cathomas R, Bernhard J, Kotrubczik NM, D'Addario G, Pilop C, Weber DC, Bodis S, Pless M, Mayer M, Stupp R. Outcome, quality of life and cognitive function of patients with brain metastases from non-small cell lung cancer treated with whole brain radiotherapy combined with gefitinib or temozolomide. A randomised phase II trial of the Swiss Group for Clinical Cancer Research (SAKK 70/03). Eur J Cancer. 2012 Feb;48(3):377-84. doi: 10.1016/j.ejca.2011.10.016. Epub 2011 Nov 15. PMID 22093943
- [Background] Haie-Meder C, Pellae-Cosset B, Laplanche A, Lagrange JL, Tuchais C, Nogues C, Arriagada R. Results of a randomized clinical trial comparing two radiation schedules in the palliative treatment of brain metastases. Radiother Oncol. 1993 Feb;26(2):111-6. doi: 10.1016/0167-8140(93)90091-l. PMID 7681997
- [Background] Davey P, Hoegler D, Ennis M, Smith J. A phase III study of accelerated versus conventional hypofractionated whole brain irradiation in patients of good performance status with brain metastases not suitable for surgical excision. Radiother Oncol. 2008 Aug;88(2):173-6. doi: 10.1016/j.radonc.2008.05.020. Epub 2008 Jun 12. PMID 18555546
- [Background] Rades D, Kieckebusch S, Lohynska R, Veninga T, Stalpers LJ, Dunst J, Schild SE. Reduction of overall treatment time in patients irradiated for more than three brain metastases. Int J Radiat Oncol Biol Phys. 2007 Dec 1;69(5):1509-13. doi: 10.1016/j.ijrobp.2007.05.014. Epub 2007 Aug 6. PMID 17689033
- [Background] Hendriks LE, Troost EG, Steward A, Bootsma GP, De Jaeger K, van den Borne BE, Dingemans AM. Patient selection for whole brain radiotherapy (WBRT) in a large lung cancer cohort: Impact of a new Dutch guideline on brain metastases. Acta Oncol. 2014 Jul;53(7):945-51. doi: 10.3109/0284186X.2014.906746. Epub 2014 Apr 23. PMID 24754845
- [Background] El Gantery MM, Abd El Baky HM, El Hossieny HA, Mahmoud M, Youssef O. Management of brain metastases with stereotactic radiosurgery alone versus whole brain irradiation alone versus both. Radiat Oncol. 2014 May 20;9:116. doi: 10.1186/1748-717X-9-116. PMID 24884624
- [Background] Kondziolka D, Patel A, Lunsford LD, Kassam A, Flickinger JC. Stereotactic radiosurgery plus whole brain radiotherapy versus radiotherapy alone for patients with multiple brain metastases. Int J Radiat Oncol Biol Phys. 1999 Sep 1;45(2):427-34. doi: 10.1016/s0360-3016(99)00198-4. PMID 10487566
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Background] Frazier JL, Batra S, Kapor S, Vellimana A, Gandhi R, Carson KA, Shokek O, Lim M, Kleinberg L, Rigamonti D. Stereotactic radiosurgery in the management of brain metastases: an institutional retrospective analysis of survival. Int J Radiat Oncol Biol Phys. 2010 Apr;76(5):1486-92. doi: 10.1016/j.ijrobp.2009.03.028. Epub 2009 Jul 18. PMID 19619958
- [Background] Bhatnagar AK, Flickinger JC, Kondziolka D, Lunsford LD. Stereotactic radiosurgery for four or more intracranial metastases. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):898-903. doi: 10.1016/j.ijrobp.2005.08.035. Epub 2005 Dec 9. PMID 16338097
- [Background] Serizawa T, Iuchi T, Ono J, Saeki N, Osato K, Odaki M, Ushikubo O, Hirai S, Sato M, Matsuda S. Gamma knife treatment for multiple metastatic brain tumors compared with whole-brain radiation therapy. J Neurosurg. 2000 Dec;93 Suppl 3:32-6. doi: 10.3171/jns.2000.93.supplement. PMID 11143259
- [Background] Park SH, Hwang SK, Kang DH, Lee SH, Park J, Hwang JH, Hamm IS, Park YM. Gamma knife radiosurgery for multiple brain metastases from lung cancer. J Clin Neurosci. 2009 May;16(5):626-9. doi: 10.1016/j.jocn.2008.08.003. Epub 2009 Mar 5. PMID 19268596
- [Background] Raldow AC, Chiang VL, Knisely JP, Yu JB. Survival and intracranial control of patients with 5 or more brain metastases treated with gamma knife stereotactic radiosurgery. Am J Clin Oncol. 2013 Oct;36(5):486-90. doi: 10.1097/COC.0b013e31825494ef. PMID 22706180
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Shaw E, Scott C, Souhami L, Dinapoli R, Kline R, Loeffler J, Farnan N. Single dose radiosurgical treatment of recurrent previously irradiated primary brain tumors and brain metastases: final report of RTOG protocol 90-05. Int J Radiat Oncol Biol Phys. 2000 May 1;47(2):291-8. doi: 10.1016/s0360-3016(99)00507-6. PMID 10802351
- [Background] Blonigen BJ, Steinmetz RD, Levin L, Lamba MA, Warnick RE, Breneman JC. Irradiated volume as a predictor of brain radionecrosis after linear accelerator stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):996-1001. doi: 10.1016/j.ijrobp.2009.06.006. Epub 2009 Sep 23. PMID 19783374
- [Background] Minniti G, Clarke E, Lanzetta G, Osti MF, Trasimeni G, Bozzao A, Romano A, Enrici RM. Stereotactic radiosurgery for brain metastases: analysis of outcome and risk of brain radionecrosis. Radiat Oncol. 2011 May 15;6:48. doi: 10.1186/1748-717X-6-48. PMID 21575163
- [Background] Bauman G, Yartsev S, Fisher B, Kron T, Laperriere N, Heydarian M, VanDyk J. Simultaneous infield boost with helical tomotherapy for patients with 1 to 3 brain metastases. Am J Clin Oncol. 2007 Feb;30(1):38-44. doi: 10.1097/01.coc.0000245473.41035.c4. PMID 17278893
- [Background] Lagerwaard FJ, van der Hoorn EA, Verbakel WF, Haasbeek CJ, Slotman BJ, Senan S. Whole-brain radiotherapy with simultaneous integrated boost to multiple brain metastases using volumetric modulated arc therapy. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):253-9. doi: 10.1016/j.ijrobp.2009.03.029. Epub 2009 Jul 4. PMID 19577856
- [Background] Edwards AA, Keggin E, Plowman PN. The developing role for intensity-modulated radiation therapy (IMRT) in the non-surgical treatment of brain metastases. Br J Radiol. 2010 Feb;83(986):133-6. doi: 10.1259/bjr/28596848. Epub 2009 Dec 17. PMID 20019176
- [Background] Meany HJ, Fox E, McCully C, Tucker C, Balis FM. The plasma and cerebrospinal fluid pharmacokinetics of erlotinib and its active metabolite (OSI-420) after intravenous administration of erlotinib in non-human primates. Cancer Chemother Pharmacol. 2008 Aug;62(3):387-92. doi: 10.1007/s00280-007-0616-3. Epub 2007 Oct 12. PMID 17932674
- [Background] Wang M, Jing Z, Mingjiang C. Cerebral penetration of gefitinib in patients with lung adenocarcinoma[J]. J Clin Oncol, 2011, 29(suppl); abstr7608
- [Background] Togashi Y, Masago K, Fukudo M, Tsuchido Y, Okuda C, Kim YH, Ikemi Y, Sakamori Y, Mio T, Katsura T, Mishima M. Efficacy of increased-dose erlotinib for central nervous system metastases in non-small cell lung cancer patients with epidermal growth factor receptor mutation. Cancer Chemother Pharmacol. 2011 Oct;68(4):1089-92. doi: 10.1007/s00280-011-1691-z. Epub 2011 Jun 17. PMID 21681573
- [Background] Togashi Y, Masago K, Masuda S, Mizuno T, Fukudo M, Ikemi Y, Sakamori Y, Nagai H, Kim YH, Katsura T, Mishima M. Cerebrospinal fluid concentration of gefitinib and erlotinib in patients with non-small cell lung cancer. Cancer Chemother Pharmacol. 2012 Sep;70(3):399-405. doi: 10.1007/s00280-012-1929-4. Epub 2012 Jul 18. PMID 22806307
- [Background] Wu YL, Zhou C, Cheng Y, Lu S, Chen GY, Huang C, Huang YS, Yan HH, Ren S, Liu Y, Yang JJ. Erlotinib as second-line treatment in patients with advanced non-small-cell lung cancer and asymptomatic brain metastases: a phase II study (CTONG-0803). Ann Oncol. 2013 Apr;24(4):993-9. doi: 10.1093/annonc/mds529. Epub 2012 Nov 4. PMID 23129122
- [Background] Park SJ, Kim HT, Lee DH, Kim KP, Kim SW, Suh C, Lee JS. Efficacy of epidermal growth factor receptor tyrosine kinase inhibitors for brain metastasis in non-small cell lung cancer patients harboring either exon 19 or 21 mutation. Lung Cancer. 2012 Sep;77(3):556-60. doi: 10.1016/j.lungcan.2012.05.092. Epub 2012 Jun 5. PMID 22677429
- [Background] Porta R, Sanchez-Torres JM, Paz-Ares L, Massuti B, Reguart N, Mayo C, Lianes P, Queralt C, Guillem V, Salinas P, Catot S, Isla D, Pradas A, Gurpide A, de Castro J, Polo E, Puig T, Taron M, Colomer R, Rosell R. Brain metastases from lung cancer responding to erlotinib: the importance of EGFR mutation. Eur Respir J. 2011 Mar;37(3):624-31. doi: 10.1183/09031936.00195609. Epub 2010 Jul 1. PMID 20595147
- [Background] Barsukov VS. [Quantitative description of the process of radiation inactivation of cells. VIII. Microdosimetry in the analysis of the reproductive death of eukaryotic cells]. Tsitologiia. 1977 Sep;19(9):991-9. Russian. PMID 929699
- [Background] Tanaka T, Munshi A, Brooks C, Liu J, Hobbs ML, Meyn RE. Gefitinib radiosensitizes non-small cell lung cancer cells by suppressing cellular DNA repair capacity. Clin Cancer Res. 2008 Feb 15;14(4):1266-73. doi: 10.1158/1078-0432.CCR-07-1606. PMID 18281562
- [Background] Chinnaiyan P, Huang S, Vallabhaneni G, Armstrong E, Varambally S, Tomlins SA, Chinnaiyan AM, Harari PM. Mechanisms of enhanced radiation response following epidermal growth factor receptor signaling inhibition by erlotinib (Tarceva). Cancer Res. 2005 Apr 15;65(8):3328-35. doi: 10.1158/0008-5472.CAN-04-3547. PMID 15833866
- [Background] Wang M, Morsbach F, Sander D, Gheorghiu L, Nanda A, Benes C, Kriegs M, Krause M, Dikomey E, Baumann M, Dahm-Daphi J, Settleman J, Willers H. EGF receptor inhibition radiosensitizes NSCLC cells by inducing senescence in cells sustaining DNA double-strand breaks. Cancer Res. 2011 Oct 1;71(19):6261-9. doi: 10.1158/0008-5472.CAN-11-0213. Epub 2011 Aug 18. PMID 21852385
- [Background] Zhuang H, Yuan Z, Wang J, Zhao L, Pang Q, Wang P. Phase II study of whole brain radiotherapy with or without erlotinib in patients with multiple brain metastases from lung adenocarcinoma. Drug Des Devel Ther. 2013 Oct 8;7:1179-86. doi: 10.2147/DDDT.S53011. eCollection 2013. PMID 24133369
- [Background] Welsh JW, Komaki R, Amini A, Munsell MF, Unger W, Allen PK, Chang JY, Wefel JS, McGovern SL, Garland LL, Chen SS, Holt J, Liao Z, Brown P, Sulman E, Heymach JV, Kim ES, Stea B. Phase II trial of erlotinib plus concurrent whole-brain radiation therapy for patients with brain metastases from non-small-cell lung cancer. J Clin Oncol. 2013 Mar 1;31(7):895-902. doi: 10.1200/JCO.2011.40.1174. Epub 2013 Jan 22. PMID 23341526